CLINICAL TRIAL: NCT06446323
Title: Comparison of Minimal Effective Dose of Sucrose for Pain Relief in Neonates After Minor Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rawalpindi Medical College (Other)
Responsible Party: Principal Investigator, Mehak Fatima, Mehak Fatima, Rawalpindi Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Rawalpindi MU
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Post Procedural Pain Management in Neonates
Keywords: sucrose solution, pain relief, neonates, minor procedure, Premature Infant Pain Profile

STUDY DESIGN:
Intervention Model Description: In this parallel interventional study, neonates who have undergone minor procedures and are admitted to the neonatal intensive care unit are randomly assigned to one of two groups: Group I or Group II. Group I receives a 0.2 ml dose of sucrose solution, while Group II receives a 0.5 ml dose.
  The study follows a parallel design, where each group receives a different intervention (different doses of sucrose solution) simultaneously. This design allows for a direct comparison between the two interventions while minimizing potential biases.
  After administration of the respective doses, the neonates are monitored for pain intensity using the Premature Infant Pain Profile (PIPP). Data on pain scores are collected and analyzed using statistical methods, such as those performed with SPSS version 25.0.
  The primary objective of this parallel interventional study is to determine which dose of sucrose solution (0.2 ml or 0.5 ml) is more effective in reducing post-procedural pain in neonates.
Who Masked: Investigator
Masking Description: The investigators responsible for assessing the primary outcome measure, pain intensity using the Premature Infant Pain Profile (PIPP), are blinded to the treatment allocation. While neonates and healthcare providers administering the interventions are aware of the treatment groups, the investigators conducting the outcome assessments remain unaware of which dose of sucrose solution each neonate received. This masking of the investigators helps mitigate potential bias in the assessment of pain relief efficacy. However, it is acknowledged that complete masking of all parties involved is not feasible due to the nature of the interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I: Neonates receiving a 0.2 ml dose of sucrose solution (Active Comparator): Participants in this arm receive a 0.2 ml dose of sucrose solution. Care providers administer the specified dose of sucrose solution to neonates who have undergone minor procedures and are experiencing post-procedural pain. The dose is administered orally, following standardized protocols. Participants in this group are monitored for pain intensity using the Premature Infant Pain Profile (PIPP) by investigators who are masked to the treatment allocation. Data on pain scores and any adverse events are recorded and analyzed as part of the study.
  Interventions: Drug: 0.2 ml dose of sucrose
- Group II: Neonates receiving a 0.5 ml dose of sucrose solution. (Active Comparator): Participants in this arm receive a 0.5 ml dose of sucrose solution. Similar to Arm 1, care providers administer the specified dose orally to neonates following minor procedures. The administration is conducted according to standardized protocols. Pain intensity in this group is also monitored using the Premature Infant Pain Profile (PIPP) by investigators who remain masked to the treatment allocation. Data collected includes pain scores and any adverse events experienced by participants.
  Interventions: Drug: 0.2 ml dose of sucrose

INTERVENTIONS:
Drug: 0.2 ml dose of sucrose — Both interventions aim to provide pain relief to neonates following minor procedures by administering sucrose solution orally. The study evaluates the efficacy of each dose (0.2 ml vs. 0.5 ml) in reducing post-procedural pain intensity, as measured by the Premature Infant Pain Profile (PIPP). Additionally, any adverse events associated with the administration of sucrose solution are documented and analyzed as part of the study.
  Other Names: 0.5 ml dose of sucrose

SUMMARY:
Type of Study: Randomized Controlled Trial Aim: To compare the effectiveness of two doses of sucrose solution for pain relief in neonates after minor procedures.

Participants' Tasks:

Receive either 0.2 ml or 0.5 ml of sucrose solution. Undergo minor procedures. Pain intensity assessment using the Premature Infant Pain Profile (PIPP).

Comparison Groups:

Researchers compared the effects of administering 0.2 ml and 0.5 ml doses of sucrose solution on post-procedural pain in neonates.

DETAILED DESCRIPTION:
This study is a randomized controlled trial conducted at the Department of Pediatric Surgery, Holy Family Hospital, Rawalpindi, from March 2023 to February 2024. It aims to compare the effectiveness of two different doses of sucrose solution (0.2 ml versus 0.5 ml) for pain relief in neonates after minor procedures.

Objective:

To compare the outcome of 0.2 ml versus 0.5 ml sucrose solution for pain relief in neonates after minor procedures.

Study Design:

Randomized Controlled Trial

Study Place and Duration:

Department of Pediatric Surgery, Holy Family Hospital, Rawalpindi, March 2023 to February 2024.

Participants and Methods:

Total of 148 neonates enrolled who underwent minor procedures and were admitted to the neonatal intensive care unit.

Randomly divided into two groups:

Group I: Administered 0.2 ml of sucrose solution Group II: Administered 0.5 ml of sucrose solution Pain intensity measured using the Premature Infant Pain Profile (PIPP). Data analyzed using SPSS version 25.0.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term neonates admitted to the neonatal intensive care unit (NICU) and high dependency unit (HDU) at the Department of Pediatric Surgery, Holy Family Hospital, Rawalpindi.

Exclusion Criteria:

* Neonates with contraindications for sucrose administration, including:

Inability to swallow. Pharmacological muscle relaxation. Heavy sedation. Neonates who are unable to clearly view the infant's face, hindering accurate pain assessment

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
pain intensity in neonates | immediately after administrating the sucrose
  The primary outcome of this study is the measurement of pain intensity in neonates following minor procedures, assessed using the Premature Infant Pain Profile (PIPP). The PIPP is a validated tool used to evaluate pain in preterm and term neonates based on behavioral and physiological indicators.

CONTACTS AND LOCATIONS:
Locations (1):
- Mehak Fatima, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR